CLINICAL TRIAL: NCT00623831
Title: A Phase 1 Study of Mixed Bacteria Vaccine (MBV) in Patients With Tumors Expressing NY-ESO-1 Antigen.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ludwig Institute for Cancer Research (Other)
Collaborators: Krankenhaus Nordwest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUD2005-003; 2006-002015-27 (EudraCT Number)
Record Dates: First submitted 2008-02-04; First posted 2008-02-26 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Melanoma; Sarcoma; Gastrointestinal Stromal Tumor (GIST); Head and Neck Cancer; Transitional Cell Carcinoma; Prostate Cancer; Ovarian Carcinoma; Esophageal Cancer; Breast Cancer
Keywords: MBV; Mixed Bacterial Vaccine; NY-ESO-1
MeSH Terms: conditions — Melanoma; Sarcoma; Gastrointestinal Stromal Tumors; Head and Neck Neoplasms; Carcinoma, Transitional Cell; Prostatic Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Subjects received MBV at a starting dose of 250 EU (dose level 1) twice weekly, with intrasubject dose escalations for each subsequent administration in the absence of a DLT until the desired pyrogenic effect was observed. The maximum possible dose to be investigated was 547,000 EU (dose level 8).
  Interventions: Biological: Mixed bacterial vaccine
- Cohort 2 (Experimental): Subjects received MBV twice weekly at the fixed dose (60,800 EU [dose level 6]) that was determined to be the pyrogenic dose level in Cohort 1.
  Interventions: Biological: Mixed bacterial vaccine

INTERVENTIONS:
Biological: Mixed bacterial vaccine — MBV was administered twice weekly by subcutaneous injection in Cohort 1 and by intralesional (preferred) or subcutaneous (if intralesional not possible) injection in Cohort 2. In Cohort 1, the MBV starting dose was 250 EU (dose level 1) with possible intrasubject escalations up to 547,000 EU (dose level 8). In Cohort 2, all subjects received MBV at a fixed dose of 60,800 EU (dose level 6).
  Other Names: MBV

SUMMARY:
This was a phase 1, open-label, multiple dose, single-arm study. The mixed bacteria vaccine (MBV) was administered at a starting dose of 250 EU (1 µL) and escalated in each subject to a dose inducing the desired pyrogenic effect, defined as a body temperature of 38°C to 39.5°C. The primary objective was to determine the safety profile of MBV in subjects with malignant tumors that expressed the NY-ESO-1 antigen and to identify the dose that induced the desired pyrogenic effect. Secondary objectives were to evaluate the immunological effects and tumor response of subjects following vaccination.

DETAILED DESCRIPTION:
Subjects in Cohort 1 were enrolled to receive MBV subcutaneously at a starting dose of 250 EU (1 µL; dose level 1) administered twice weekly. In the absence of a dose-limiting toxicity (DLT), the MBV dose was escalated in each subject to the MBV dose that elicited the desired pyrogenic effect, or up to the maximum dose of 547,000 EU (dose level 8). Once the desired pyrogenic effect was observed, subjects received MBV twice weekly for 4 doses at the pyrogenic dose level.

Subjects in Cohort 2 were enrolled to receive MBV at the pyrogenic dose level (determined to be 60,800 EU [dose level 6]) twice weekly for 6 weeks. Vaccinations were injected intralesionally if possible and subcutaneously if intralesional injection was not possible. If a fever of 39.5°C to 40°C was observed, the subject's dose was reduced to dose level 5 (20,300 EU [81 μL]).

Subjects were observed at the clinic for up to 6 hours following each vaccination, with vital signs measured hourly. At baseline and throughout the study, subjects were assessed for NY-ESO-1-specific humoral and cellular immunity, chemistry, hematology, and cytokine analysis (interleukin [IL]-1, IL-6, interferon [IFN]-γ, and tumor necrosis factor [TNF]-α). Safety was monitored continuously throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic melanoma, head and neck cancer, transitional cell carcinoma, sarcoma, gastrointestinal stroma tumor (GIST) or prostate cancer.
2. Tumor expression of NY-ESO-1 by reverse transcriptase and polymerase chain reaction (RT-PCR) analysis, preferably, or immunohistochemistry.
3. Expected survival of at least 6 months.
4. Karnofsky performance status ≥ 70%.
5. Fully recovered from surgery.
6. Declined, intolerated or completed standard therapy defined as follows for each tumor entity:

   1. Melanoma - resistance or intolerance to dacarbazine.
   2. Sarcoma - resistance or intolerance to anthracyclines and to one platinum-containing chemotherapy regimen, no indication for irradiation.
   3. GIST - failure or intolerance of imatinib and sunitinib.
   4. Head and neck cancer - no indication for irradiation, resistance or intolerance to platinum-containing chemotherapy.
   5. Transitional cell carcinoma - resistance or intolerance to cisplatin combined with gemcitabine.
   6. Prostate cancer- failure of antihormonal treatment and resistance or intolerance to docetaxel.
   7. Ovarian carcinoma - failure of standard chemotherapy consisting of a platinum agent combined with a taxane and of an anthracycline.
   8. Esophageal cancer - failure of standard chemotherapy consisting of a platinum agent.
   9. Breast cancer- failure or intolerance of standard first-, second- and third-line chemotherapy consisting of a taxane and anthracycline. No indication or resistance to standard antihormonal treatment. No indication or resistance to human epidermal growth factor receptor (HER)-2-neu targeted therapy. No indication or resistance to irradiation and/or surgery.
7. Within the last 2 weeks prior to study day 1, vital laboratory parameters must have been within the normal range, except for the following laboratory parameters, which must have been within the ranges specified:

   * Absolute neutrophil count (ANC): ≥ 1,000/mm3
   * Platelet count: ≥ 75,000/mm3
   * Alanine aminotransferase (ALT): ≤ 5 x upper limit of normal (ULN)
   * Aspartate aminotransferase (AST): ≤ 5 x ULN
   * Total bilirubin: ≤ 2.5 x ULN
   * Creatinine: ≤ 2 mg/dL
8. Age ≥ 18 years.
9. Able and willing to give written informed consent.

Exclusion Criteria:

1. Clinically significant heart disease (New York Heart Association Class III or IV).
2. Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders.
3. Subjects with serious intercurrent illness requiring hospitalization.
4. Known human immunodeficiency virus positivity.
5. Chemotherapy, radiation therapy or immunotherapy within 4 weeks prior to first dose of study agent (6 weeks for nitrosoureas).
6. Known autoimmune disease (rheumatoid arthritis, systemic lupus erythematosus), as these conditions might have interfered with the evaluation of the induced immune response. Subjects with vitiligo or melanoma-associated hypopigmentation were not excluded.
7. Chronic use of immunosuppressive drugs such as systemic corticosteroids.
8. Other malignancy within 3 years prior to entry into the study, except for treated non-melanoma skin cancer and cervical carcinoma in situ.
9. Mental impairment that may have compromised the ability to give informed consent and comply with the requirements of the study.
10. Lack of availability for immunological and clinical follow-up assessments.
11. Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study agent.
12. Pregnancy or breastfeeding.
13. Women of childbearing potential: Refusal or inability to use effective means of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elke Jager, MD, Principal Investigator — Krankenhaus Nordwest
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data have been published

REFERENCES:
- [Result] Karbach J, Neumann A, Brand K, Wahle C, Siegel E, Maeurer M, Ritter E, Tsuji T, Gnjatic S, Old LJ, Ritter G, Jager E. Phase I clinical trial of mixed bacterial vaccine (Coley's toxins) in patients with NY-ESO-1 expressing cancers: immunological effects and clinical activity. Clin Cancer Res. 2012 Oct 1;18(19):5449-59. doi: 10.1158/1078-0432.CCR-12-1116. Epub 2012 Jul 30. PMID 22847809

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Subjects received MBV twice weekly by subcutaneous injection at a starting dose of 250 EU (dose level 1), with intrasubject dose escalations for each subsequent administration in the absence of a dose-limiting toxicity (DLT) until the desired pyrogenic effect was observed.
- Cohort 2: Subjects received MBV twice weekly by intralesional (preferred) or subcutaneous (if intralesional not possible) injection at the fixed dose (60,800 EU [dose level 6]) that was determined to be the pyrogenic dose level in Cohort 1.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 13 | 4
Completed | 12 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Progressive Disease | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Enrolled Subjects
Groups:
- Cohort 1: Subjects received MBV twice weekly by subcutaneous injection at a starting dose of 250 EU (dose level 1), with intrasubject dose escalations for each subsequent administration in the absence of a DLT until the desired pyrogenic effect was observed.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 13 | 4 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 11
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (11.7) | 55.5 (11.3) | 57.4 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 4 | 13
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 4 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 13 | 4 | 17
Diagnosis at Study Entry [Count of Participants; unit: Participants]
  Melanoma | 7 | 2 | 9
  Sarcoma | 2 | 1 | 3
  Prostate cancer | 2 | 0 | 2
  Head and neck cancer | 1 | 0 | 1
  Breast cancer | 0 | 1 | 1
  Transitional cell carcinoma | 1 | 0 | 1
Stage IV Disease at Study Entry [Count of Participants; unit: Participants] | 13 | 4 | 17
Baseline Karnofsky Performance Status [Count of Participants; unit: Participants] — 100%: Normal no complaints; no evidence of disease. 90%: Able to carry on normal activity; minor signs or symptoms of disease. 80%: Normal activity with effort; some signs or symptoms of disease. 70%: Cares for self; unable to carry on normal activity or to do active work.
  Participants
    70% | 2 | 0 | 2
    80% | 4 | 0 | 4
    90% | 4 | 0 | 4
    100% | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Analysis of treatment-emergent adverse events (TEAEs) reported from clinical laboratory tests, physical examinations, and vital signs from pre-treatment through 4 weeks after the last dose of study treatment.
Time Frame: Up to 3 months
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- Cohort 1 (Safety Analysis Set): Subjects received MBV twice weekly by subcutaneous injection at a starting dose of 250 EU (dose level 1), with intrasubject dose escalations for each subsequent administration in the absence of a DLT until the desired pyrogenic effect was observed.
- Cohort 2 (Safety Analysis Set): Subjects received MBV twice weekly by intralesional (preferred) or subcutaneous (if intralesional not possible) injection at the fixed dose (60,800 EU [dose level 6]) that was determined to be the pyrogenic dose level in Cohort 1.
Arm/Group | Cohort 1 (Safety Analysis Set) | Cohort 2 (Safety Analysis Set)
Number analyzed (Participants) | 13 | 4
participants
  Any TEAE | 13 | 4
  Grade 3 TEAE | 3 | 2
  Grade 4 TEAE | 0 | 0
  Grade 5 TEAE (Death) | 1 | 0
  Treatment-related TEAE | 9 | 3
  SAE | 1 | 1
  TEAE leading to withdrawal | 0 | 0

2. Primary Outcome: Number of Participants With Pyrogenicity at Each Dose Level Tested in the Intrasubject Dose Escalation Performed Over a Dose Range of 250 to 547,000 EU
Description: Intrasubject dose escalation performed over a dose range of 250 to 547,000 EU until achievement of the desired pyrogenic effects (i.e., body temperature increase to 38°C to 39.5°C). Of note, the median pyrogenic dose was 60,800 EU.
Time Frame: Weeks 1 through 6
Population: The Safety Analysis Set comprises all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Cohort 1 (Safety Analysis Set)
Number analyzed (Participants) | 13
participants
  Pyrogenic Dose: 250 EU | 1
  Pyrogenic Dose: 750 EU | 1
  Pyrogenic Dose: 2250 EU | 1
  Pyrogenic Dose: 20,300 EU | 1
  Pyrogenic Dose: 60,800 EU | 2
  Pyrogenic Dose: 182,000 EU | 2
  Pyrogenic Dose: 547,000 EU | 3
  Desired Pyrogenic Effect Not Observed | 1
  Discontinued Before Pyrogenic Effect Observed | 1

3. Secondary Outcome: Number of Participants With Serum NY-ESO-1-specific Immune Responses
Description: Serum NY-ESO-1-specific immune responses evaluated by humoral immunity (antibodies measured by ELISA), cellular immunity (CD8+ T-cell and CD4+ T-cell measured by ELISPOT), and cytokine activation (measured by ELISA) from pre-treatment through 4 weeks after the last dose of study treatment. [Note: CD = cluster of differentiation; IFN =interferon; IL = interleukin; TNF = tumor necrosis factor]
Time Frame: Up to 3 months
Population: The Immune Response Analysis Set comprises all subjects who achieved the desired pyrogenic effects.
Measure: Number; unit: participants
Groups:
- Cohort 1 (Immune Response Analysis Set): Subjects received MBV twice weekly by subcutaneous injection at a starting dose of 250 EU (dose level 1), with intrasubject dose escalations for each subsequent administration in the absence of a DLT until the desired pyrogenic effect was observed.
Arm/Group | Cohort 1 (Immune Response Analysis Set)
Number analyzed (Participants) | 12
participants
  Antibody Sero(+) Pre- and Post-treatment | 9
  Antibody Sero(-) Pre- and Post-treatment | 2
  Antibody Sero(-) Pre-treatment, (+) Post-treatment | 1
  CD4+ Pre- and Post-treatment | 5
  CD4- Pre- and Post-treatment | 6
  CD4 Not Evaluable | 1
  CD8+ Pre- and Post-treatment | 7
  CD8- Pre- and Post-treatment | 5
  Increase of ≥ 2 Cytokines Post-treatment | 11
  IL-6 Increase Post-treatment | 11
  TNF-α Increase Post-treatment | 5
  IFN-γ Increase Post-treatment | 5
  IL-2 Increase Post-treatment | 3
  IL-Iβ Increase Post-treatment | 2
  IL-8 Increase Post-treatment | 2
  IL-10 Increase Post-treatment | 2
  IL-12 Increase Post-treatment | 1
  IL-5 Increase Post-treatment | 0

4. Secondary Outcome: Number of Participants With Best Overall Tumor Response
Description: Tumor responses evaluated using computed tomography and categorized according to RECIST version 1.0 at pre-treatment and 4 weeks after the last dose of study treatment. Per RECIST v1.0 for target lesions and assessed by MRI: Complete Response (CR): Disappearance of all target lesions [no evidence of disease]; Partial Response (PR): ≥ 30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD): ≥ 20% increase in the sum of the longest diameter of target lesions; Stable Disease (SD): small changes that do not meet above criteria.
Time Frame: Up to 3 months
Population: The Tumor Response Analysis Set comprises all subjects who had an end-of-study tumor assessment performed.
Measure: Number; unit: participants
Groups:
- Cohort 1 (Tumor Response Analysis Set): Subjects received MBV twice weekly by subcutaneous injection at a starting dose of 250 EU (dose level 1), with intrasubject dose escalations for each subsequent administration in the absence of a DLT until the desired pyrogenic effect was observed.
- Cohort 2 (Tumor Response Analysis Set): Subjects received MBV twice weekly by intralesional (preferred) or subcutaneous (if intralesional not possible) injection at the fixed dose (60,800 EU [dose level 6]) that was determined to be the pyrogenic dose level in Cohort 1.
Arm/Group | Cohort 1 (Tumor Response Analysis Set) | Cohort 2 (Tumor Response Analysis Set)
Number analyzed (Participants) | 12 | 3
participants
  No evidence of disease | 2 | 1
  Partial response | 1 | 0
  Stable disease | 0 | 1
  Progressive disease | 9 | 1

ADVERSE EVENTS:
Time Frame: All AEs occurring between the signing of informed consent and the off-study date were documented, regardless of the causal relationship to study drug. AEs occurring after the first dose of study drug were considered treatment emergent (i.e., TEAEs). The AE reporting period for this study was up to 3 months for each subject.
Description: AE documentation included onset/resolution dates, severity using NCI CTCAE (v3.0), seriousness, study drug action taken, treatment, and outcome. In summaries, treatment-related AEs included those with a "possible", "probable", or "definite" relationship to study drug; preferred terms were counted only once per subject at the maximum reported grade.
Arm/Group | Cohort 1 | Cohort 2
Serious Adverse Events (participants affected / at risk) | 1/13 | 1/4
Other Adverse Events (participants affected / at risk) | 13/13 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2 (N=4)
Rapid disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Grade 5; not related to study drug
Increased pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Grade 3; not related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=13) | Cohort 2 (N=4)
Pain at injection site (General disorders) | 4 | 2
CRP elevation (Investigations) | 3 | 2
Edema (General disorders) | 4 | 0
Weakness (General disorders) | 2 | 2
Chills (General disorders) | 1 | 2
Fever (General disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Tachycardia (Cardiac disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Fatigue (General disorders) | 1 | 1
Flu-like feeling (General disorders) | 1 | 1
Increased dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Abrasion head (General disorders) | 0 | 1
Angina tonsillaris (General disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder pressure (Renal and urinary disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Candida infection urine (Renal and urinary disorders) | 1 | 0
Co-reaction of prior injection sites (General disorders) | 0 | 1
Common cold (Infections and infestations) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Decubitus (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Expectoration (General disorders) | 1 | 0
Feeling of pressure in head (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0
Hematoma due to fall (by accident) (Injury, poisoning and procedural complications) | 1 | 0
Herpes labialis (Infections and infestations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Inappetence (Metabolism and nutrition disorders) | 1 | 0
Increased pain (General disorders) | 1 | 0
Increased swollen tongue (Gastrointestinal disorders) | 1 | 0
Increased visual disturbance (Eye disorders) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infection at peg (Infections and infestations) | 1 | 0
Mucositis (General disorders) | 1 | 0
Pain (intermittent; face/head/tongue) (General disorders) | 1 | 0
Pain at scar (General disorders) | 1 | 0
Pain limbs (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain right leg (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain upper abdomen (Gastrointestinal disorders) | 1 | 0
Pruritus at injection site (Skin and subcutaneous tissue disorders) | 1 | 0
Reddening at port catheter site (Skin and subcutaneous tissue disorders) | 1 | 0
Reduced performance status (General disorders) | 1 | 0
Reduced perfusion in toes (Vascular disorders) | 1 | 0
Soft stool (Gastrointestinal disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Subjective feeling of sickness (General disorders) | 1 | 0
Suspected candidosis glans penis (Infections and infestations) | 1 | 0
Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Symptomatic ascites (Gastrointestinal disorders) | 1 | 0
Thoracic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombosis (pelvic) (Vascular disorders) | 1 | 0
Thrush to the mouth (Infections and infestations) | 0 | 1
Tickle in throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tumor-related thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Wound eye (Eye disorders) | 1 | 0
Increased pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less